CLINICAL TRIAL: NCT04686370
Title: Effect of Different Implant Surface Treatments on Bony Changes Around Mandibular Implants for Completely Edentulous Patients (A Split-mouth Comparative Study)
Brief Title: Effect of Different Implant Surface Treatments on Bony Changes Around Mandibular Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwan Mohamed Abdelsalam, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-2-34
Record Dates: First submitted 2020-11-25; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Complete Edentulism
Keywords: Dental implant; Surface treatment; Laser; Sandblasted Acid-etched implants; Delayed-loading; Bony changes; Marginal bone loss

STUDY DESIGN:
Intervention Model Description: one single group will receive both types of dental implants (Split-mouth)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sandblasted acid-etched implants (Active Comparator): implant will be installed intraforaminal
  Interventions: Other: laser treated implant surface
- laser treated implants (Experimental): implant will be installed intraforaminal
  Interventions: Other: laser treated implant surface

INTERVENTIONS:
Other: laser treated implant surface — Better marginal bone stability is expected for this type

SUMMARY:
The research will be conducted to report which type of surface treatment of dental implants that can be successful and aids in increasing bone to implant contact and how it affects the bony changes around the implants installed in mandibular arches for completely edentulous patients or whether there are specific precautions to be taken into consideration during implant planning concerned with the type of surface microstructure treatment and recommendations needed.

DETAILED DESCRIPTION:
Primary objective:

PICO P: Completely edentulous patients I: Laser surface treatment of implants C: Sandblasted Acid etched surface treatment O: Bony changes

Each Participants will have 2 implants;one laser surface treated implants and another sandblasted acid-etched implant (split-mouth) installed in the intra-foraminal area of mandibular arch prosthetically driven by the prepared conventional denture. MS and AF are responsible for delayed-loading of the denture and will measure bony changes around laser treated surface implants using radiographic assessment using long paralleling technique periapical digital x-ray(SOREDEX™ DIGORA™ Optime)

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients
* Angle's class 1 skeletal relationship
* Normal facial asymmetry
* Cooperative patients
* Adequate inter-arch spcae not less than 12mm

Exclusion Criteria:

* Tempromandibular joint disorder
* Uncontrolled diabetes
* Bleeding disorders or anticoagulant therapy
* Flabby tissues or sharp mandibular residual ridge
* Heavy smoker
* Patient's with neuromuscular disorders
* Patients on chemotherapy or radiotherapy
* Severe psychiatric disorders

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Marginal bone stability around dental implants | 1 year
  Measuring amount of marginal bone loss by radiographic assessment using long paralleling technique periapical digital x-ray(SOREDEX™ DIGORA™ Optime)

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Mohamed, Investigator, Principal Investigator — Cairo University
Locations (1):
- Faculty of dentistry,cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No